CLINICAL TRIAL: NCT01738490
Title: Long-term Stability and Survival Rates of a Novel Oticon Medical Bone Conduction Device Implant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oticon Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C33
Record Dates: First submitted 2012-11-28; First posted 2012-11-30 (Estimated); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Deafness; Hearing Loss; Hearing Loss, Conductive; Hearing Disorders; Ear Diseases; Otorhinolaryngologic Diseases
Keywords: Bone anchored hearing aid; Bone anchored implant; Implant stability; Wide diameter implant; Linear incision; Ponto
MeSH Terms: conditions — Deafness; Hearing Loss; Hearing Loss, Conductive; Hearing Disorders; Ear Diseases; Otorhinolaryngologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wide diameter implant (Other): Bone anchored hearing implant For the wide diameter arm (test group), the Ponto wide implant (diameter 4,5mm, length 4mm) and abutment 6mm developed by Oticon Medical AB (Gothenburg, Sweden) will be installed.
  Interventions: Device: Bone anchored hearing implant
- Control group (Other): Bone anchored hearing implant For the control group, the previous generation Ponto implant (diameter 3,75mm, length 4mm) and 6mm abutment (Oticon Medical AB, Gothenburg, Sweden) will be installed.
  Interventions: Device: Bone anchored hearing implant

INTERVENTIONS:
Device: Bone anchored hearing implant
  Other Names: Ponto implant; Bone anchored hearing aid

SUMMARY:
The overall aim of the study is to investigate the Ponto wide implant considering; initial implant stability, stability over time, skin reaction and long term success when loaded at 3 weeks post surgery. Patients' quality of life improvements following implantation will also be surveyed.

More specifically the primary objective of this clinical study is to test the hypothesis

* The new Ponto wide diameter implant offers increased implant stability measured as ISQ (implant stability quotient) compared to the previous generation Ponto implant.

And the secondary objective is to

* Investigate when in time implant stability is the lowest as the initial mechanical stability is gradually replaced by biological stability

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Patient indicated for an ear level bone anchored sound processor
* Bone thickness at the implant site of at least 4 mm

Exclusion Criteria:

* Longer abutment (>6mm) required
* Inability to participate in follow-up
* Psychiatric disease in the medical history
* Mental disability
* Presumed doubt, for any reason, that the patient will be able to show up on all follow ups
* Diseases or treatments known to compromise the bone quality at the implant site, e.g. radiotherapy, osteoporosis, diabetes mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2012-06; Primary Completion 2014-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
ISQ (Implant Stability Quotient) | Surgery (0 days)
  ISQ (implant Stability Quotient) is a measurement scale for use with the Resonance Frequency Analysis (RFA) method of determining implant stability. The measurement is made using the Osstell Mentor equipment (Osstell, Sweden) with SmartPegs. ISQ values range from 1 to 100, the higher the score the higher the stability. The highest and lowest score obtained from perpendicular measurements will be registered.
ISQ (Implant Stability Quotient) | 7 days after surgery
ISQ (Implant Stability Quotient) | 14 days after surgery
ISQ (Implant Stability Quotient) | 21 days after surgery
ISQ (Implant Stability Quotient) | 28 days after surgery
ISQ (Implant Stability Quotient) | 6 weeks after surgery
ISQ (Implant Stability Quotient) | 12 weeks after surgery
ISQ (Implant Stability Quotient) | 6 months after surgery
ISQ (Implant Stability Quotient) | 12 months after surgery
ISQ (Implant Stability Quotient) | 24 months after surgery
ISQ (Implant Stability Quotient) | 36 months after surgery

SECONDARY OUTCOMES:
Time of minimum ISQ (Implant stability quotient) | 0, 7, 14, 21 and 28 days after surgery
  Implant stability can be seen as a combination of mechanical stability, which is the result of compressed bone holding the implant tightly in place, and biological stability, which is the result of new bone forming at the site of implantation and osseointegration. Mechanical stability is generally high immediately after implant placement and is decreasing with time. Biological stability, on the other hand, is non-existent immediately after placement and increases with time. The final stability level for an implant is the sum of the two. There is likely to be an initial decrease in stability followed by a subsequent increase as the implant becomes biologically stable. ISQ (implant Stability Quotient) is a measurement scale for use with the Resonance Frequency Analysis (RFA) method of determining implant stability.
ISQ (Implant stability quotient) gradient | 0, 7, 14, 21 and 28 days, 6 weeks, 12weeks, 6 months after surgery
  ISQ (implant stability quotient) per time unit gives a measure of osseointegration speed.
Skin condition according to Holgers score | 7 days after surgery
  Holgers score is a standardized scale to clinically assess skin condition around a percutaneous implant
Skin condition according to Holgers score | 14 days after surgery
Skin condition according to Holgers score | 21 days after surgery
Skin condition according to Holgers score | 28 days after surgery
Skin condition according to Holgers score | 6 weeks after surgery
Skin condition according to Holgers score | 12 weeks after surgery
Skin condition according to Holgers score | 6 months after surgery
Skin condition according to Holgers score | 12 months after surgery
Skin condition according to Holgers score | 24 months after surgery
Skin condition according to Holgers score | 36 months after surgery
Glasgow Benefit Inventory Questionnaire | 3 months after surgery
  Glasgow Benefit Inventory Questionnaire (GBI) 18-item, post-surgical questionnaire given to patients. The GBI measures the change in health status produced by surgical interventions (here, "health status" is the general perception of well-being, including total psychological, social, and physical well being).
Glasgow Benefit Inventory Questionnaire | 12 months after surgery
Abbreviated Profile of Hearing Aid Benefit (APHAB) questionnaire | Before surgery
  The APHAB is a 24-item self-assessment inventory in which patients report the amount of trouble they are having with communication or noises in various everyday situations. Benefit is calculated by comparing the patient's reported difficulty in the unaided condition with their amount of difficulty when using amplification. The APHAB produces scores for 4 subscales: Ease of Communication (EC), Reverberation (RV), Background Noise (BN), and Aversiveness (AV).
Abbreviated Profile of Hearing Aid Benefit (APHAB) questionnaire | 6 months after surgery
Abbreviated Profile of Hearing Aid Benefit (APHAB) questionnaire | 36 months after surgery
Glasgow Health Status Inventory (GHSI) questionnaire | Before surgery
  The Glasgow Health Status Inventory is an 18 item questionnaire. It assesses health state, by measuring the effect of a health problem on the quality of life of a person. It allows cross-comparison among many health conditions, among different health interventions, and among demographic and cultural subgroups.
Glasgow Health Status Inventory (GHSI) questionnaire | 6 months after surgery
Glasgow Health Status Inventory (GHSI) questionnaire | 36 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Myrthe KS Hol, MD, PhD, Principal Investigator — University Medical Center St Radboud, Nijmegen, The Netherlands
Locations (1):
- University Medical Center St Radboud, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nelissen RC, den Besten CA, Mylanus EA, Hol MK. Stability, survival, and tolerability of a 4.5-mm-wide bone-anchored hearing implant: 6-month data from a randomized controlled clinical trial. Eur Arch Otorhinolaryngol. 2016 Jan;273(1):105-11. doi: 10.1007/s00405-015-3593-x. Epub 2015 Mar 20. PMID 25790770